CLINICAL TRIAL: NCT02719405
Title: A Prospective Randomized Controlled Trial to Evaluate the Effect of Infant Formula on the Resolution of Cow's Milk Allergy of Infancy
Brief Title: Impact of Infant Formula on Resolution of Cow's Milk Allergy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mead Johnson Nutrition (Industry)
Responsible Party: Principal Investigator, Wayne G. Shreffler, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2015P000962
Record Dates: First submitted 2015-10-30; First posted 2016-03-25 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Milk Allergy
Keywords: milk; allergy; tolerance
MeSH Terms: conditions — Milk Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amino Acid Formula (Placebo Comparator)
  Interventions: Dietary Supplement: Amino Acid Formula
- EHCF (Active Comparator): Extensively Hydrolyzed Casein Formula
  Interventions: Dietary Supplement: Extensively Hydrolyzed Casein Formula
- EHCF + LGG (Active Comparator): Extensively Hydrolyzed Casein Formula + Lactobacillus GG
  Interventions: Dietary Supplement: Lactobacillus GG; Dietary Supplement: Extensively Hydrolyzed Casein Formula

INTERVENTIONS:
Dietary Supplement: Lactobacillus GG — Lactobacillus GG
  Arms: EHCF + LGG
Dietary Supplement: Extensively Hydrolyzed Casein Formula — Extensively Hydrolyzed Casein Formula
  Arms: EHCF; EHCF + LGG
Dietary Supplement: Amino Acid Formula — Amino Acid Formula
  Arms: Amino Acid Formula

SUMMARY:
Primary Endpoint

-The percentage of subjects who develop tolerance to cow's milk protein by 12 months post randomization to study formula.

Secondary Endpoints

* Tolerance

  * The transcriptional profile of milk-specific T cells by clinical outcome.
  * Growth and Weight Velocity
  * Stool Consistency and Frequency
  * The estimated frequency of milk-specific T cells by clinical outcome.
  * The TCR diversity of milk-specific T cells by clinical outcome.
  * The milk allergen component-specific IgE, IgG4 and IgA by clinical outcome.
* Safety

  * The rate of reported adverse events by treatment group.

DETAILED DESCRIPTION:
Cow's Milk Allergy (CMA) is prevalent and most often presents during infancy. Disease manifestations vary through a range of immediate and delayed inflammatory responses to milk protein from anaphylaxis to enterocolitis. The natural history is also highly variable; most children will achieve clinical tolerance early in life, while a minority will have disease persisting to adulthood for reasons that are not known. Most presentations are mild and are managed by restriction or reduction of immunologically intact milk protein with reintroduction sometime after a year of age; however, there are data to suggest that some level of antigenic stimulation may be beneficial. Furthermore, recent data suggest that oral probiotic exposure may also promote tolerance, though the kinetics of tolerance acquisition, the interaction between these two factors (probiotics and milk antigen exposure) and their relationship to regulatory T cell responses are all poorly defined. Therefore, there is an unmet need to identify dietary interventions, along with corresponding immune responses, that favor the promotion of tolerance.

A major objective will be to measure the effect probiotics have on the development of tolerance to milk antigen over time. By following these infants during the first year of life, and repeatedly collecting blood and stool samples from them, we will be poised to analyze their stool microbiome signatures, and we will estimate the frequency, phenotype and TCR diversity of milk-specific T cells over time. By repeatedly challenging them with more immunologically intact milk protein, we will better define the kinetics of CMA resolution and its association to these variables. This information is likely to further elucidate CMA disease mechanisms and identify possible biomarkers of disease resolution versus persistence. It will be directly useful for evaluating the efficacy of probiotics and hydrolyzed formula for promoting milk tolerance.

ELIGIBILITY:
Inclusion Criteria (to consent):

* Infants 0-120 days of age with suspected CMA, as determined by the pediatrician or specialist, will be referred to the study. A Standard Operating Procedures (SOP) document will be provided for the clinicians to help guide their referral to the study. Physician diagnosis of CMA will be based on the following:
* Physician documented, gross or persistent microscopic blood in stool (3 positive guaiac cards on three separate stools) in the absence of other explanation (e.g., fissure, moderate-to-severe constipation) AND / OR

Infant with at least one gastrointestinal, dermatological, or respiratory allergic manifestation suggestive of CMA:

* Gastrointestinal: Chronic Diarrhea, Constipation or Vomiting/Gastro-esophageal reflux
* Dermatologic: Atopic Dermatitis or Urticaria
* Respiratory: Cough, Allergic rhinitis or Recurrent Wheezing
* General:Colic / Irritability
* No change in treatment with medications during the 7 days preceding the elimination diet and no expected change in medications during the DBPCFCs (unless otherwise medically necessary)
* Signed informed consent obtained for infants participation in the study
* Signed authorization obtained to use and/or disclose Protected Health Information for infant from birth through the length of the study period
* Willingness to comply with following inclusion criteria if found to have a positive DBPCFC screen:

  1. Caregiver(s) agree to comply with the infant elimination diet given to them by the investigator for the duration of the study
  2. Mother agrees to follow an elimination diet throughout duration of breast feeding
  3. Parent(s) or legally authorized representative agrees not to enroll infant in another interventional clinical study while participating in this study

Inclusion Criteria (to randomization):

* Positive Double Blind Placebo Controlled Food Challenge (DBPCFC).

Exclusion Criteria (to consent):

* History of anaphylaxis to milk
* Use of probiotics
* Use in the previous 4 weeks of systemic steroids
* Use of systemic immunomodulatory treatment, including biologics with an immune target such as Xolair
* Known eosinophilic GI disorders
* Episode(s) of severe repetitive vomiting and lethargy prompting an emergency room visit and occurring within 4 hours of ingesting a milk protein (i.e. consistent with FPIES)
* Co-existing autoimmune or other chronic disease or serious health problem, including celiac disease, inflammatory bowel disease, malignancy, congenital, metabolic or genetic disorders or malformations
* Intention to exclusively breast feed
* Infants born at less than 36 weeks gestation (35 weeks + 6 days is considered 35 weeks gestation)

Exclusion Criteria (to randomization):

* Severe reaction to Milk Protein during the DBPCFC

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects who develop tolerance to cow's milk protein by 12 months post randomization to study formula. | 12 months post randomization

SECONDARY OUTCOMES:
Safety as assessed by adverse events graded using the NCI-CTCAE scale by treatment group. | 36 months
  The rate of reported adverse events by treatment group.
Tolerance as assessed by the transcriptional profile of milk-specific T cells by clinical outcome. | 36 months
Tolerance as assessed by weight for age Z-scores. | 36 months
Tolerance as assessed by length for age Z-scores. | 36 months
Tolerance as assessed by weight for length Z-scores. | 36 months
Tolerance as assessed by stool consistency using the Bristol Stool Chart. | 36 months
Tolerance as assessed by stool frequency. | 36 months
Tolerance as assessed by changes in the stool microbiome. | 36 months
Tolerance as assessed by the estimated frequency of milk-specific T cells by clinical outcome. | 36 months
Tolerance as assessed by the TCR diversity of milk-specific T cells by clinical outcome. | 36 months
Tolerance as assessed by the milk allergen component-specific IgE, IgG4 and IgA by clinical outcome. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Wayne G Shreffler, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Woburn Pediatric Associates, Woburn, Massachusetts

REFERENCES:
- [Derived] Amari S, Shahrook S, Namba F, Ota E, Mori R. Branched-chain amino acid supplementation for improving growth and development in term and preterm neonates. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD012273. doi: 10.1002/14651858.CD012273.pub2. PMID 33006765